CLINICAL TRIAL: NCT07401706
Title: Effects of Vestibular Rehabilitation in Comparison With Routine Physical Therapy on Stability, Kinesiophobia and Return to Sports in Athletes With Post Concussion Syndrome
Brief Title: Effects of Vestibular Rehabilitation and Routine Physical Therapy in Athletes With Post Concussion Syndrome
Acronym: PCS BESS IPRRS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lahore University of Biological and Applied Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DPT/ERB/25; Syeda Farwa Aitbar (Registry Identifier: U1111-1333-2730)
Record Dates: First submitted 2026-02-03; First posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Post Concussion Syndrome
Keywords: TAMPA; BESS; IPRRS; RPT; Athletes; Post concussion syndrome; vestibular rehabilitation; stability; kinesiophobia; return to sports
MeSH Terms: conditions — Post-Concussion Syndrome; Kinesiophobia

STUDY DESIGN:
Intervention Model Description: not needed
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vestibular Rehabilitation (Experimental): The experimental group received a structured Vestibular Rehabilitation Program that included balance training, habituation exercises, and gaze stabilization exercises. These interventions were designed to improve postural stability, reduce dizziness and motion sensitivity, and enhance visual vestibular interaction. Each session lasted 30 minutes, was conducted three times per week, and continued for a total of four weeks under the supervision of a licensed physical therapist.
  Interventions: Other: Intervention 1
- Routine Physical Therapy (Active Comparator): The control group received Routine Physical Therapy, consisting of ankle strategy exercises to improve postural control through ankle musculature and coordination, along with elliptical training at sub-symptom threshold levels to promote aerobic conditioning. Similar to the experimental group, these sessions were performed for 30 minutes, three times per week, for four weeks, and were supervised by a licensed physical therapist.
  Interventions: Other: Control Arm (Conventional Therapy)

INTERVENTIONS:
Other: Intervention 1 — Vestibular Rehabilitation includes balance training, habituation exercises, and gaze stabilization/oculomotor training. Balance training is performed 3 times per week, with intensity progressed from static stance to dynamic tasks such as foam beam and head turns. The time is three sets each for 30 seconds, making a total treatment time of 30 minutes. The type of balance training includes static balance (single-leg and tandem) and dynamic balance (foam beam walking with head turns). Habituation exercises were performed three times per week, with intensity of three sets of 100 feet distance covered while gradually increasing complexity from head turns to ball toss. The time is 3 minute activity performed following 1 minute rest, making a total treatment time of 30 minutes. The type of exercise includes VOR habituation such as head turn with ambulation, ball toss up and down while walking, and ball toss side to side while walking. Gaze stabilization/oculomotor training is also performed t
  Arms: Vestibular Rehabilitation
Other: Control Arm (Conventional Therapy) — Routine Physical Therapy consist of ankle strategies and elliptical training. Ankle strategies are performed three times per week with intensity progressed from rocker board to dual-task activities. The time duration is three sets of two minutes with two minutes of rest, resulting in a total treatment time of 30 minutes. The type of exercise involves rocker board movements in anterior/posterior and medial/lateral directions, with or without ball toss or gaze fixation (X1 viewing). Elliptical training is also performed three times per week at mild exertion, starting at level 1 and with asymptomatic threshold. Each session includes a 5-minute warm-up, 20 minutes of training, and a 5-minute cool-down, making the total treatment time 30 minutes. The mode of exercise is submaximal aerobic exercise on an elliptical trainer
  Arms: Routine Physical Therapy

SUMMARY:
This randomized controlled trial with a parallel design was conducted over six months at Ghurki Trust Teaching Hospital to compare the effects of Vestibular Rehabilitation and Routine Physical Therapy on stability, kinesiophobia, and return to sports in athletes with post-concussion syndrome. A total of 34 participants aged 12 to 30 years were enrolled based on specific diagnostic criteria. Non probability convenient sampling was used, followed by random allocation into experimental and control groups through computer generated sequencing and sealed envelope concealment. Single blinding was done, with participants unaware of their assigned intervention.

The experimental group received a Vestibular Rehabilitation program consisting of balance training, habituation exercises, and gaze stabilization, while the control group underwent Routine Physical Therapy involving ankle strategies and elliptical training. Both interventions were administered for 30 minutes, three times per week, over four weeks. Outcomes were measured pre- and post-intervention using validated tools: the Balance Error Scoring System (BESS) for postural stability, the Urdu version of the Tampa Scale of Kinesiophobia (TSK), and the Injury Psychological Readiness to Return to Sport Scale (I-PRRS). Data analysis was performed using SPSS version 26, employing appropriate parametric or non-parametric tests based on normality, with significance set at p < 0.05. Ethical approval was obtained, informed consent was secured, and all procedures adhered to established ethical standards.

ELIGIBILITY:
Inclusion Criteria:

1. Age 12 to 30 years
2. Fulfil the criteria of post concussion syndrome as highlighted by Tator et al.(2016)which requires presence of at least 3 or more persistent symptoms from standardized list
3. Sustained a mTBI in past 3 to 12 weeks
4. Having ongoing symptoms from list in PCSS that started 72 hrs or less after an impact
5. Exhibit objective deficits on standardized baseline examination enabling vestibular and ocular dysfunction

Exclusion Criteria:

* Have a chronic infectious disease.

  * Uncontrolled hypertension.
  * Other neurological disorders (not attributed to their primary diagnosis).
  * Cancer treatment (other than basal cell carcinoma), craniotomy, or refractory subdural hematoma.
  * Those on long term use of psychoactive drugs that compromise their ability to perform study activities
  * Those with pacemakers or elevated cardiovascular risk.
  * Ongoing litigation surrounding their injury.
  * Have been diagnosed with a severe brain injury prior to enrollment, or their post concussive symptoms have persisted beyond 12

Ages: 12 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 34 (Estimated)
Dates: Start 2026-03-22 (Estimated); Primary Completion 2026-06-22 (Estimated); Study Completion 2026-07-22 (Estimated)

PRIMARY OUTCOMES:
Kinesiophobia | 4 weeks
  For kinesiophobia the Urdu version of Tampa scale was used to asses athletes. The Urdu version of the TSK is considered to be a valid and reliable tool for assessing kinesiophobia.
  1. = strongly disagree
  2. = disagree
  3. = agree
  4. = strongly agree Tampa Scale for Kinesiophobia (TSK) The TSK is a self report questionnaire used to measure fear of movement.
  It contains 17 items, each scored on a 4-point Likert scale:
  Total score range: 17 to 68 Reverse scored items: 4, 8, 12, 16 (For these items: 1↔4, 2↔3)
Stability | 4 weeks
  The Balance Error Scoring System (BESS) has demonstrated excellent validity and reliability in patients. Test-retest reliability was strong, with ICC values ranging from 0.88 to 0.99 (average 0.90) and Cronbach's alpha between 0.90 and 0.99, indicating high internal consistency.Types of Errors
  Hands lifted off the iliac crest
  Opening eyes
  Step, stumble, or fall
  Moving hip into >30° abduction
  Lifting forefoot or heel
  Remaining out of the test position for more than 5 seconds
  The BESS is calculated by adding one error point for each error during the six 20-second tests.
  Which Foot Was Tested
  * Left
  * Right (i.e., the non-dominant foot)
  Score Card (Number of Errors) Test Condition Firm Surface Foam Surface Double-Leg Stance (feet together) Single-Leg Stance (non-dominant foot) Tandem Stance (non-dominant foot in back)
  Total Scores:
  BESS Total:60
Return to sports | 4 weeks
  The Injury Psychological Readiness to Return to Sport (I-PRRS) scale was selected as it has undergone translation and validation in Dutch athletes. The instrument demonstrated strong internal consistency (Cronbach's α = 0.94) and excellent test-retest reliability (ICC = 0.89).
  0 = no confidence at all, 50 = moderate confidence, 100 = complete confidence. Rate Value My overall confidence to play is ________ My confidence to play without pain is ________ My confidence to give 100 percent effort is ________ My confidence to not concentrate on the injury is ________ My confidence in the injured body part to handle the demands of the situation is ________ My confidence in my skill level/ability is ________
  Total: ________

CONTACTS AND LOCATIONS:
Overall Officials: Tariq Shafi, Study Chair — Lahore University of Biological And Applied Health Sciences; Syeda Farwa Aitbar, DPT, Principal Investigator — Lahore College of Physical Therapy; Maheen Mazhar, DPT, Principal Investigator — Lahore College of Physical Therapy; Ayesha Naeem Khan, DPT, Principal Investigator — Lahore College of Physical Therapy

IPD SHARING:
Plan to Share IPD: Yes
After the publication
Supporting Information: Study Protocol, SAP
Time Frame: June 2026-October 2026